CLINICAL TRIAL: NCT03973619
Title: Urethral Stricture Repair: A Prospective Randomized Analysis Between Jugal or Labial Graft in Buccal Mucosa Urethroplasty
Brief Title: Urethral Stricture: A Comparison Between Jugal or Labial Graft Urethroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Rafael Carvalho Ipe da Silva, Principal Investigator, MD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170319
Record Dates: First submitted 2019-05-15; First posted 2019-06-04 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Urethral Stricture
Keywords: urethral stricture; mucosa graft; jugal graft,; labial graft; success rate
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labial (Active Comparator): Patients who received a labial graft as replacement of urethral tissue
  Interventions: Procedure: Labial Graft
- Jugal (Active Comparator): Patients who received a jugal (inner cheek) graft as replacement of urethral tissue
  Interventions: Procedure: Jugal Graft

INTERVENTIONS:
Procedure: Labial Graft — As replacement of the damaged urethral tissue, we used a buccal mucosa graft (labial graft).
  Arms: Labial
Procedure: Jugal Graft — As replacement of the damaged urethral tissue, we used a buccal mucosa graft(inner cheek - jugal graft).
  Arms: Jugal

SUMMARY:
Buccal mucosa urethroplasty is a current fashion in urethral stricture management. In our university centre (Hospital de Clínicas de Porto Alegre) is a common surgical treatment choice. This paper aims to evaluate the success rate of this treatment after randomized choice between labial and jugal (inner cheek) grafts during the past two years.

DETAILED DESCRIPTION:
Free dorsal graft urethroplasty, first described by Barbagli et al, has been shown better results than ventral grafts. Fixed grafts on the corpora cavernosa results in a better mechanical support and vascular supply, with less chance to complications such as pseudodiverticula and sacculations either a better urethral phisiology.

This study aims to evaluate the current surgical management in our centre: buccal mucosa graft urethroplasty with jugal or labial replacement, comparing their group success rate and complications between the groups in patients led to surgery from October 2016 to June 2018.

Prospective analysis from urethral stricture surgical HCPA patient data by dorsal buccal mucosa graft urethroplasty. The graft choice were done by a software. Longer stricture with transoperative need for the two grafts use were excluded. Success rate were measured with a no stricture de novo or absence of complications in a six month interval.

ELIGIBILITY:
Inclusion Criteria:

* Urethral Stricture Diagnosis
* Indication for buccal mucosa graft urethroplasty
* Accept the Informed Consent Term (patient or responsible)

Exclusion Criteria:

* Severe urethral stricture which a two-staged procedure are required
* Long strictures which need a both types of buccal mucosa graft due its length.
* Refuse to ICT for the patient ou it responsible

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Overall Success Rate | 6 months
  Absence of surgical intervention after prior surgery
Labial Group Success Rate | 6 months
  Absence of surgical intervention after prior surgery on patients who received a labial graft.
Jugal Group Success Rate | 6 months
  Absence of surgical intervention after prior surgery on patients who received a inner cheek graft.
Latex Catheter Success Rate | 6 months
  Absence of surgical intervention on patients who used a latex catheter indwelling after prior surgery.
Silicon Catheter Success Rate | 6 months
  Absence of surgical intervention on patients who used a silicon catheter indwelling after prior surgery.

SECONDARY OUTCOMES:
Stricture Etiology | 24 months
  Evaluation of the etiology of the stricture (trauma, other, infectious) on patients included on Labial and Jugal Groups
Stricture Localization | 24 months
  Evaluation of the stricture localization (penile, bulbar/bulbomembranous or combined) on patients included on Labial and Jugal Groups
Stricture Size | 24 months
  Evaluation of the stricture length (cm) on patients included on Labial and Jugal Groups
Demographic Data | 24 months
  Evaluation of the demographic data relationship with the results (age, cystotomy, cystostomy time, tobacco use, diabetes, balanitis xerotica, UTI infection, serum creatin levels) included on Labial and Jugal groups

CONTACTS AND LOCATIONS:
Overall Officials: Brasil S Neto, Phd MD, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbagli G, Palminteri E, Guazzoni G, Montorsi F, Turini D, Lazzeri M. Bulbar urethroplasty using buccal mucosa grafts placed on the ventral, dorsal or lateral surface of the urethra: are results affected by the surgical technique? J Urol. 2005 Sep;174(3):955-7; discussion 957-8. doi: 10.1097/01.ju.0000169422.46721.d7. PMID 16094007
- [Background] Bracka A. A versatile two-stage hypospadias repair. Br J Plast Surg. 1995 Sep;48(6):345-52. doi: 10.1016/s0007-1226(95)90023-3. PMID 7551506
- [Background] Morey AF, McAninch JW. When and how to use buccal mucosal grafts in adult bulbar urethroplasty. Urology. 1996 Aug;48(2):194-8. doi: 10.1016/S0090-4295(96)00154-9. PMID 8753728
- [Background] Palminteri E, Lumen N, Berdondini E, Di Pierro GB, Cucchiarale G, Tenti G, De Nunzio C. Two-sided dorsal plus ventral oral graft bulbar urethroplasty: long-term results and predictive factors. Urology. 2015 Apr;85(4):942-7. doi: 10.1016/j.urology.2015.01.013. PMID 25817122
- [Background] Pansadoro V, Emiliozzi P, Gaffi M, Scarpone P, DePaula F, Pizzo M. Buccal mucosa urethroplasty in the treatment of bulbar urethral strictures. Urology. 2003 May;61(5):1008-10. doi: 10.1016/s0090-4295(02)02585-2. PMID 12736025
- [Background] Sharma AK, Chandrashekar R, Keshavamurthy R, Nelvigi GG, Kamath AJ, Sharma S, Venkatesh GK. Lingual versus buccal mucosa graft urethroplasty for anterior urethral stricture: a prospective comparative analysis. Int J Urol. 2013 Dec;20(12):1199-203. doi: 10.1111/iju.12158. Epub 2013 Apr 21. PMID 23601029
- [Background] Barbagli G, Palminteri E, Lazzeri M, Guazzoni G, Turini D. Long-term outcome of urethroplasty after failed urethrotomy versus primary repair. J Urol. 2001 Jun;165(6 Pt 1):1918-9. doi: 10.1097/00005392-200106000-00018. PMID 11371881
- [Background] Martinez-Pineiro JA, Martinez-Pineiro L, Tabernero A. [Substitution urethroplasties with free graft buccal mucosa]. Arch Esp Urol. 1998 Sep;51(7):645-59. Spanish. PMID 9807890
- [Background] Barbagli G, Pellegrini G, Corradini F, Montorsi F, Sansalone S, Butnaru D, Lazzeri M. One-stage Penile Urethroplasty Using Oral Mucosal Graft and Glue. Eur Urol. 2016 Dec;70(6):1069-1075. doi: 10.1016/j.eururo.2016.04.025. Epub 2016 May 6. PMID 27160949
- [Background] Aldaqadossi H, El Gamal S, El-Nadey M, El Gamal O, Radwan M, Gaber M. Dorsal onlay (Barbagli technique) versus dorsal inlay (Asopa technique) buccal mucosal graft urethroplasty for anterior urethral stricture: a prospective randomized study. Int J Urol. 2014 Feb;21(2):185-8. doi: 10.1111/iju.12235. Epub 2013 Aug 12. PMID 23931150
- [Background] Fichtner J, Filipas D, Fisch M, Hohenfellner R, Thuroff JW. Long-term outcome of ventral buccal mucosa onlay graft urethroplasty for urethral stricture repair. Urology. 2004 Oct;64(4):648-50. doi: 10.1016/j.urology.2004.05.011. PMID 15491691
- [Background] Asopa HS, Garg M, Singhal GG, Singh L, Asopa J, Nischal A. Dorsal free graft urethroplasty for urethral stricture by ventral sagittal urethrotomy approach. Urology. 2001 Nov;58(5):657-9. doi: 10.1016/s0090-4295(01)01377-2. PMID 11711331
- [Background] Akyuz M, Gunes M, Koca O, Sertkaya Z, Kanberoglu H, Karaman MI. Evaluation of intraoral complications of buccal mucosa graft in augmentation urethroplasty. Turk J Urol. 2014 Sep;40(3):156-60. doi: 10.5152/tud.2014.46343. PMID 26328170
- [Background] Barbagli G, Vallasciani S, Romano G, Fabbri F, Guazzoni G, Lazzeri M. Morbidity of oral mucosa graft harvesting from a single cheek. Eur Urol. 2010 Jul;58(1):33-41. doi: 10.1016/j.eururo.2010.01.012. Epub 2010 Jan 19. PMID 20106587
- [Background] Elbaz J, Le Long E, Dugardin F, Sibert L, Peron JM. [Buccal mucosal graft for the treatment of urethral stricture]. Ann Chir Plast Esthet. 2012 Dec;57(6):626-9. doi: 10.1016/j.anplas.2010.09.008. Epub 2010 Oct 14. French. PMID 20950921